CLINICAL TRIAL: NCT05724212
Title: Evaluation of a CD4/CD8+ Interferon Gamma Release Assay for Monitoring Anti-Tuberculosis Treatment
Acronym: IGRA/MAT-1
Status: Active, not recruiting | Type: Observational
Sponsor: Paola Mantegani (Other)
Responsible Party: Sponsor-Investigator, Paola Mantegani, Research manager, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: IGRA/MAT-1
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Interferon-gamma Release Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Control Group (healthy subject)
  Interventions: Diagnostic Test: Interferon gamma release assay (IGRA)
- Subject with Pulmonary Tuberculosis (PTB)
  Interventions: Diagnostic Test: Interferon gamma release assay (IGRA)

INTERVENTIONS:
Diagnostic Test: Interferon gamma release assay (IGRA) — in vitro test

SUMMARY:
Evaluate the possibility of using an IGRA (Interferon-γ Release Assay) test for monitoring the response to anti-tuberculosis therapy by studying the correlation between the variation in the Interferon-gamma (IFN-γ) response to the QFT-Plus test in the two tubes containing antigens and the gold standard for monitoring TB therapy (culture conversion) in patients with slide positive/culture positive and slide negative/culture positive PTB.

Evaluate the level of agreement between the results of the new QFT Access test and the results of the QFT plus and culture in patients diagnosed with active tuberculosis. To evaluate the level of agreement between QFT Access test results and QFT Plus results in healthy controls and contacts.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms consistent with a high probability of having PULMONARY TB disease (probable case), such that they are receiving or are likely to receive ther-apy for active PTB (therapy must not have been initiated for more than 72 hours before recruitment into the study).
2. Positive sputum smear for AAR
3. Positive culture for mycobacterium tuberculosis (confirmed PTB case).
4. Positive nucleic acid amplification (NAA) test for mycobacterium tuberculosis.

Exclusion Criteria:

1. Taken therapy for active tuberculosis or latent TB infection for more than 72 hours.
2. Culture confirmation of M. tuberculosis not obtained.
3. Age less than 18 years.
4. Immunosuppression: HIV-infection, solid organ transplantation, stem cell transplantation, rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: San Raffaele Hospital wards
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of a CD4/CD8+ Interferon Gamma Release Assay for monitoring anti-Tuberculosis treatment | 1. At time of diagnosis (t0) 2. 30+ 4 days after anti-TB treatment initiation (t1) 3. 2 months after anti-TB treatment initiation (t2) 4. At the end of the anti-TB therapy (6 to 9 months) (t3)
  Define the degree of correlation between changes in IFN-γ response in the first antigen tube (TB1) and the newly added antigen tube (TB2) and the reference stand-ard of treatment response (culture conversion) in smear-positive and smear-negative/culture-positive pulmonary TB cases

CONTACTS AND LOCATIONS:
Overall Officials: Daniela M Cirillo, MD,PhD, Principal Investigator — IRCCS San Raffaele Scientific Institute Via Olgettina 60 20132 Milan Italy
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy